CLINICAL TRIAL: NCT01791153
Title: A Phase III, Multicenter, Randomized, Double-Blind Placebo-Controlled Study to Assess the Efficacy and Safety of Tocilizumab in Subjects With Giant Cell Arteritis
Brief Title: An Efficacy and Safety Study of Tocilizumab (RoActemra/Actemra) in Participants With Giant Cell Arteritis (GCA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA28119; 2011-006022-25 (EudraCT Number)
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — tocilizumab; Prednisone; Adrenal Cortex Hormones; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part 1: Tocilizumab qw + 26 weeks prednisone taper (Experimental): Participants will receive tocilizumab at a dose of 162 milligrams (mg) as subcutaneous (SC) injection qw up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants will receive prednisone tapering oral daily doses during the first 26 weeks and prednisone placebo from Week 26 up to Week 52.
  Interventions: Drug: Tocilizumab; Drug: Prednisone; Drug: Prednisone Placebo
- Part 1: Tocilizumab q2w + 26 weeks prednisone taper (Experimental): Participants will receive tocilizumab at a dose of 162 mg as SC injection q2w (and tocilizumab placebo q2w starting from Week 2) up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants will receive prednisone tapering oral daily doses during the first 26 weeks and prednisone placebo from Week 26 up to Week 52.
  Interventions: Drug: Tocilizumab; Drug: Prednisone; Drug: Tocilizumab Placebo; Drug: Prednisone Placebo
- Part 1: Placebo + 26 weeks prednisone taper (Placebo Comparator): Participants will receive tocilizumab placebo as SC injection qw up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants will receive prednisone tapering oral daily doses during the first 26 weeks and prednisone placebo from Week 26 up to Week 52.
  Interventions: Drug: Prednisone; Drug: Tocilizumab Placebo; Drug: Prednisone Placebo
- Part 1: Placebo + 52 weeks prednisone taper (Placebo Comparator): Participants will receive tocilizumab placebo as SC injection qw up to 52 weeks along with prednisone and/or prednisone placebo according to a protocol-defined schedule. Participants will receive prednisone tapering oral daily doses for 52 weeks.
  Interventions: Drug: Prednisone; Drug: Tocilizumab Placebo; Drug: Prednisone Placebo
- Part 2: Open-Label Tocilizumab qw (Experimental): Participants without sustained remission at Week 52 will receive open-label tocilizumab at a dose of 162 mg as SC injection qw and/or corticosteroids and/or methotrexate at the discretion of the investigator for a maximum of 104 weeks.
  Interventions: Drug: Tocilizumab; Drug: Corticosteroids; Drug: Methotrexate

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered at a dose of 162 mg as SC injection qw or q2w for 52 weeks in Part 1 of the study and at a dose 162 mg as SC injection qw for 104 week at the discretion of the investigator in Part 2 of the study.
  Other Names: RoActemra, Actemra, RO4877533
  Arms: Part 1: Tocilizumab q2w + 26 weeks prednisone taper; Part 1: Tocilizumab qw + 26 weeks prednisone taper; Part 2: Open-Label Tocilizumab qw
Drug: Prednisone — Prednisone will be administered at tapering oral doses as tablets daily for 26 or 52 weeks according to the protocol-defined schedule in Part 1 of the study. Prednisone will also be administered as escape therapy to treat disease flares in an open-label manner during Part 1 at a dose and duration selected by the investigator.
  Arms: Part 1: Placebo + 26 weeks prednisone taper; Part 1: Placebo + 52 weeks prednisone taper; Part 1: Tocilizumab q2w + 26 weeks prednisone taper; Part 1: Tocilizumab qw + 26 weeks prednisone taper
Drug: Tocilizumab Placebo — Tocilizumab placebo will be administered as SC injection qw or q2w for 52 weeks in Part 1 of the study.
  Arms: Part 1: Placebo + 26 weeks prednisone taper; Part 1: Placebo + 52 weeks prednisone taper; Part 1: Tocilizumab q2w + 26 weeks prednisone taper
Drug: Prednisone Placebo — Prednisone placebo will be administered as tablets orally daily according to the protocol-defined schedule (from Week 26 to Week 52) in Part 1 of the study.
  Arms: Part 1: Placebo + 26 weeks prednisone taper; Part 1: Placebo + 52 weeks prednisone taper; Part 1: Tocilizumab q2w + 26 weeks prednisone taper; Part 1: Tocilizumab qw + 26 weeks prednisone taper
Drug: Corticosteroids — Participants without sustained remission at Week 52 will receive corticosteroids at a dose and schedule at the discretion of the investigator for a maximum of 104 weeks.
  Arms: Part 2: Open-Label Tocilizumab qw
Drug: Methotrexate — Participants without sustained remission at Week 52 will receive methotrexate at a dose and schedule at the discretion of the investigator for a maximum of 104 weeks.
  Arms: Part 2: Open-Label Tocilizumab qw

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy and safety of tocilizumab in participants with GCA. The study will consist of 2 parts: a 52-week double-blind treatment period (Part 1) followed by a 104-week open label long-term follow-up period (Part 2). In Part 1 of the study eligible participants will be randomized to receive either tocilizumab every week (qw) or every 2 weeks (q2w) or placebo for 52 weeks, with tapering oral daily doses of prednisone. After Week 52, participants in remission will stop study treatment and enter long-term follow-up, whereas participants with disease activity or flares will receive open-label tocilizumab or other treatment at the discretion of the investigator for a maximum period of 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GCA classified according to age >/=50 years; history of ESR >/=50 mm/hr or history of CRP >/=2.45 mg/dL; and at least one of the following: unequivocal cranial symptoms of GCA or symptoms of polymyalgia rheumatica [PMR]; and at least one of the following: temporal artery biopsy revealing features of GCA or evidence of large-vessel vasculitis by angiography or cross-sectional imaging
* New onset (diagnosis within 6 weeks of baseline) or refractory (diagnosis greater than [>] 6 weeks before baseline and previous treatment with >/= 40 milligrams per day prednisone [or equivalent] for at least 2 consecutive weeks at any time) GCA
* Active disease (presence of clinical signs and symptoms [cranial or PMR] and ESR >/=30 mm/hour or CRP >/=1 mg/dL) within 6 weeks of baseline visit

Exclusion Criteria:

* Major surgery within 8 weeks prior to screening or planned within 12 months after randomization
* Transplanted organs (except corneas with transplant performed >3 months prior to screening)
* Major ischemic event, unrelated to GCA, within 12 weeks of screening
* Prior treatment with any of the following: investigational agent within 12 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening; cell-depleting therapies including investigational agent; intravenous (IV) gamma globulin or plasmapheresis within 6 months of baseline; alkylating agents or with total lymphoid irradiation; tocilizumab; hydroxychloroquine, cyclosporine A, azathioprine, or mycophenolate mofetil within 4 weeks of baseline; etanercept within 2 weeks of baseline; infliximab, certolizumab, golimumab, abatacept, or adalimumab within 8 weeks of baseline; anakinra within 1 week of baseline; tofacitinib; cyclophosphamide within 6 months of baseline; >100 milligrams of daily IV methylprednisolone within 6 weeks of baseline
* Participants requiring systemic glucocorticoids for conditions other than GCA, which, in the opinion of the investigator, would interfere with adherence to the fixed glucocorticoid taper regimen and/or to assessment of efficacy in response to the test article
* History of severe allergic reactions to monoclonal antibodies or to prednisone
* Evidence of serious uncontrolled concomitant disease (for example, cardiovascular, respiratory, renal, endocrine, psychiatric, corneal ulcers/injuries, or gastrointestinal [GI] disease)
* Current liver disease, as determined by the investigator
* History of diverticulitis, inflammatory bowel disease, or other symptomatic GI tract condition that might predispose to bowel perforation
* Known active or history of recurrent bacterial, viral fungal, mycobacterial, or other infection
* Primary or secondary immunodeficiency
* Evidence of malignancies diagnosed within previous 5 years (except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that have been excised and cured)
* Inadequate hematologic, renal or liver function
* Positive for hepatitis B or hepatitis C infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2013-07-22 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (78):
- United States (14):
  - Univ of Calif., Los Angeles; Rheumatology, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rheumatology Assoc. of S. Florida - Clinical Research Center, Boca Raton, Florida
  - Sarasota Arthritis Res Center, Sarasota, Florida
  - Four Rivers Clinical Research Inc., Paducah, Kentucky
  - Rheumatology Associates, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hospital For Special Surgery; Dept of Medicine - Rheumatology, New York, New York
  - Asheville Arthritis & Osteoporosis Center, PA, Asheville, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah; Division of Rheumatology, Salt Lake City, Utah
  - Marshfield Clinic Wausau Ctr, Wausau, Wisconsin
- Belgium (2):
  - Hospital Erasme, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Clin. de Rhumatologie, Trois-Rivières, Quebec, Canada
- Nordsjællands Hospital - Hillerød;Department of Rheumatology 0731, Hillerød, Denmark
- France (6):
  - Hopital Avicenne; Medecine Interne H5, Bobigny
  - Hopital La Cavale Blanche; Rhumatologie, Brest
  - Hopital Claude Huriez; Internal Medicine, Lille
  - Hôpital de la Conception, Marseille
  - Hopital Emile Muller; Medecine Interne, Mulhouse
  - Hopital Cochin; Medecine Interne, Paris
- Germany (14):
  - Asklepios Kllinikum Bad Abbach; Klinik für Rheumatologie und Klinische Immunologie, Bad Abbach
  - Rheuma-Klinikum Bad Bramstedt Klinik fuer Rheumatologie und Immunologie, Bad Bramstedt
  - Charité Campus Mitte, Med.Klinik, Rheumatologie und Klinische Immunologie, Berlin
  - Schlosspark Klinik; Abt. Rheumatologie, Berlin
  - Universitätsklinikum "Carl Gustav Carus"; Medizinische Klinik III, Dresden
  - Universitätsklinikum Erlangen; Medizinische Klinik 3; Rheumatologie und Immunologie, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Zentrum Innere Medizin Abt.Klinische Immunologie und Rheumatologie, Hanover
  - Rheumazentrum-Ruhrgebiet, St. Josefs-Krankenhaus; Rheumatologie, Herne
  - Universitätsklinikum Jena; Klinik für Innere Medizin III, Jena
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Medizinische Klinik, Pneumologie, Mainz
  - Klinikum der Universitat Munchen; Bereich Pettenkoferstr; Rheumaeinheit der medizinischen Klinik IV, München
  - Kreiskliniken Esslingen gGmbH Klinik Plochingen Medizinische Klinik, Plochingen
  - Universitätsklinikum Tübingen Medizinische UNI-Klinik und Poliklinik Abt. Innere Medizin II, Tübingen
- Italy (7):
  - Arcispedale Santa Maria Nuova; Reumatologia, Reggio Emilia, Emilia-Romagna
  - Policlinico Univ. Uni Degli Sudi Di Udine; Clinica Di Reumatologia, Udine, Friuli Venezia Giulia
  - Università Degli Studi Di Genova - Dimi; Reumatologia, Genoa, Liguria
  - Irccs San Raffele; Div Med Gen Immunologia Clinica, Milan, Lombardy
  - A.O. Universitaria Pisana; Psichiatria, Pisa, Tuscany
  - Azienda Ospedaliera di Padova; Cattedra e Divisione di Reumatologia, Padua, Veneto
  - Azienda Ospedaliera di Verona-Ospedale Civile Maggiore, Verona, Veneto
- Netherlands (5):
  - VU Medisch Centrum; Reumatologie 4-A-A2, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Universitair Medisch Centrum Groningen, Groningen
  - Ziekenhuisgroep Twente, Hengelo, Hengelo
  - Akademisch Ziekenhuis St. Radboud; Rheumatology, Nijmegen
- Norway (3):
  - Ålesund sjukehus, Ålesund
  - Sørlandet Sykehus Kristiansand, Kristiansand
  - Rikshospitalet; Revmatologisk Avd Seksjon Barnerevmatologi, Oslo
- Poland (2):
  - Szpital Uniwersytecki; nr 2 im. Dr J. Biziela, Bydgoszcz
  - Klinika Reumatologii I Chorób Wewn. Pum W Szczecinie; Samodzielny Publiczny Szpital Kliniczny Nr 1, Szczecin
- Hospital Geral de Santo Antonio; Servico de Imunologia Clinica, Porto, Portugal
- Spain (5):
  - Hospital Univ A Coruna; Rheumatology, A Coruña, LA Coruña
  - Hospital Universitario de Canarias;servicio de Reumatologia, San Cristóbal de La Laguna, Tenerife
  - Hospital de Basurto; Servicio de Reumatologia, Bilbao, Vizcaya
  - Hospital Universitari de Bellvitge; Servicio de Reumatologia, Barcelona
  - University of Barcelona; Dept. of Internal Medicine,, Barcelona
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skånes Universitetssjukhus, Lund
  - Skånes Universitetssjukhus Malmö; Reumatologkliniken, Malmo
  - Karolinska Sjukhuset; Reumatologkliniken D2-1, Stockholm
  - Akademiska Sjukhuset; Lungmedicinska Kliniken, Uppsala
- United Kingdom (12):
  - Aberdeen Royal Infirmary; Medical Oncology Dept, Aberdeen
  - Barnsley General Hospital; Rheumatology, Barnsley
  - Old Queen Elizabeth Hospital; Pharmacy Building;Clinical Research offices, Birmingham
  - Colchester General Hospital; Aseptic Dept, Pharmacy Support Unit, Colchester, Essex
  - University of Edinburgh; The Queens Medical Research Institute, Edinburgh
  - CHAPEL ALLERTON HOSPITAL; Unit of Musculoskeletal Disease, Leeds
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Freeman Hospital; Dept of Rheumatology, Newcastle upon Tyne
  - Queen's Hospital, Romford
  - Haywood Hospital; Staffordshire Rheumatology Centre, Stoke-on-Trent
  - Royal Cornwall Hospital; Rhuematololgy Dept, Truro
  - Southend Hospital; Rheumatology Department, Westcliffe-on-sea

REFERENCES:
- [Derived] Stone JH, Han J, Aringer M, Blockmans D, Brouwer E, Cid MC, Dasgupta B, Rech J, Salvarani C, Spiera R, Unizony SH, Bao M; GiACTA investigators. Long-term effect of tocilizumab in patients with giant cell arteritis: open-label extension phase of the Giant Cell Arteritis Actemra (GiACTA) trial. Lancet Rheumatol. 2021 May;3(5):e328-e336. doi: 10.1016/S2665-9913(21)00038-2. Epub 2021 Mar 19. PMID 38279390
- [Derived] Stone JH, Spotswood H, Unizony SH, Aringer M, Blockmans D, Brouwer E, Cid MC, Dasgupta B, Rech J, Salvarani C, Spiera R, Bao M. New-onset versus relapsing giant cell arteritis treated with tocilizumab: 3-year results from a randomized controlled trial and extension. Rheumatology (Oxford). 2022 Jul 6;61(7):2915-2922. doi: 10.1093/rheumatology/keab780. PMID 34718434
- [Derived] Unizony SH, Bao M, Han J, Luder Y, Pavlov A, Stone JH. Treatment failure in giant cell arteritis. Ann Rheum Dis. 2021 Nov;80(11):1467-1474. doi: 10.1136/annrheumdis-2021-220347. Epub 2021 May 28. PMID 34049857
- [Derived] Stone JH, Tuckwell K, Dimonaco S, Klearman M, Aringer M, Blockmans D, Brouwer E, Cid MC, Dasgupta B, Rech J, Salvarani C, Schulze-Koops H, Schett G, Spiera R, Unizony SH, Collinson N. Glucocorticoid Dosages and Acute-Phase Reactant Levels at Giant Cell Arteritis Flare in a Randomized Trial of Tocilizumab. Arthritis Rheumatol. 2019 Aug;71(8):1329-1338. doi: 10.1002/art.40876. Epub 2019 Jul 3. PMID 30835950
- [Derived] Strand V, Dimonaco S, Tuckwell K, Klearman M, Collinson N, Stone JH. Health-related quality of life in patients with giant cell arteritis treated with tocilizumab in a phase 3 randomised controlled trial. Arthritis Res Ther. 2019 Feb 20;21(1):64. doi: 10.1186/s13075-019-1837-7. PMID 30786937
- [Derived] Stone JH, Tuckwell K, Dimonaco S, Klearman M, Aringer M, Blockmans D, Brouwer E, Cid MC, Dasgupta B, Rech J, Salvarani C, Schett G, Schulze-Koops H, Spiera R, Unizony SH, Collinson N. Trial of Tocilizumab in Giant-Cell Arteritis. N Engl J Med. 2017 Jul 27;377(4):317-328. doi: 10.1056/NEJMoa1613849. PMID 28745999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consists of 2 parts: a 52-week double-blind treatment period (Part 1) followed by a 104-week open label long-term follow-up period (Part 2).
Pre-assignment Details: Of the 363 participants screened, a total of 251 participants were randomized into the study. One participant who was randomized to the "Tocilizumab q2w + 26 weeks prednisone taper" group withdrew on the same day of randomization and did not receive any study treatment. This participant was not included in any of the study analyses.
Groups:
- Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper: Participants received tocilizumab at a dose of 162 milligrams (mg) as subcutaneous (SC) injection every week (qw) up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone placebo from Week 26 up to Week 52.
- Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper: Participants received tocilizumab at a dose of 162 mg as SC injection every 2 weeks (q2w) (and tocilizumab placebo q2w starting from Week 2) up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone placebo from Week 26 up to Week 52.
- Part 1: Placebo + 26 Weeks Prednisone Taper: Participants received tocilizumab placebo as SC injection qw up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone placebo from Week 26 up to Week 52.
- Part 1: Placebo + 52 Weeks Prednisone Taper: Participants received tocilizumab placebo as SC injection qw up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses for 52 weeks.
- Part 2: No Tocilizumab (Placebo in Part 1): Participants did not receive tocilizumab in Part 2 from Week 52 up to Week 156. These participants received placebo during Part 1 (Weeks 1 to 52).
- Part 2: No Tocilizumab (Tocilizumab in Part 1): Participants did not receive tocilizumab in Part 2 from Week 52 up to Week 156. These participants received tocilizumab during Part 1 (Weeks 1 to 52).
- Part 2: Tocilizumab (Placebo in Part 1): Participants received open-label tocilizumab as determined by the investigator during Part 2 of the study (from Week 52 up to Week 156). These participants received placebo during Part 1 (Weeks 1 to 52).
- Part 2: Tocilizumab (Tocilizumab in Part 1): Participants received open-label tocilizumab as determined by the investigator during Part 2 of the study (from Week 52 up to Week 156). These participants received tocilizumab during Part 1 (Weeks 1 to 52).
Period: Part 1: Blinded Period
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper | Part 2: No Tocilizumab (Placebo in Part 1) | Part 2: No Tocilizumab (Tocilizumab in Part 1) | Part 2: Tocilizumab (Placebo in Part 1) | Part 2: Tocilizumab (Tocilizumab in Part 1)
Started | 100 | 49 | 50 | 51 | 0 | 0 | 0 | 0
Completed | 85 (Completed Study to Week 52) | 41 (Completed Study to Week 52) | 44 (Completed Study to Week 52) | 46 (Completed Study to Week 52) | 0 | 0 | 0 | 0
Not Completed | 15 | 8 | 6 | 5 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 3 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Non-Compliance | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Period: Part 2: Open-label Period
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper | Part 2: No Tocilizumab (Placebo in Part 1) | Part 2: No Tocilizumab (Tocilizumab in Part 1) | Part 2: Tocilizumab (Placebo in Part 1) | Part 2: Tocilizumab (Tocilizumab in Part 1)
Started | 0 | 0 | 0 | 0 | 40 | 58 | 50 | 67
Completed | 0 | 0 | 0 | 0 | 38 | 54 | 44 | 61
Not Completed | 0 | 0 | 0 | 0 | 2 | 4 | 6 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one administration of study drug and provided at least one post-dose safety assessment.
Groups:
- Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper: Participants received tocilizumab at a dose of 162 mg as SC injection qw up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone placebo from Week 26 up to Week 52.
- Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper: Participants received tocilizumab at a dose of 162 mg as SC injection q2w (and tocilizumab placebo q2w starting from Week 2) up to 52 weeks along with prednisone and/or prednisone placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 26 weeks and prednisone placebo from Week 26 up to Week 52.
- Total: Total of all reporting groups
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper | Total
Number analyzed (Participants) | 100 | 49 | 50 | 51 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (8.50) | 69.4 (8.29) | 69.3 (8.14) | 67.8 (7.70) | 69.1 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 34 | 38 | 37 | 187
  Male | 22 | 15 | 12 | 14 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Sustained Remission at Week 52 (Tocilizumab + 26 Weeks Prednisone Taper Versus Placebo + 26 Weeks Prednisone Taper)
Description: Remission was defined as the absence of flare and normalization of the C-reactive protein (CRP) (less than [<] 1 milligram per deciliter [mg/dL]). Sustained remission was defined as the absence of flare following induction of remission within 12 weeks of randomization and maintained up to Week 52. Flare was determined by the investigator and was defined as the recurrence of signs or symptoms of GCA and/or erythrocyte sedimentation rate (ESR) greater than or equal to (>/=) 30 millimeters per hour (mm/hr) attributable to GCA. A single CRP elevation (>/=1 mg/dL) was not considered as a sign of flare, unless the CRP remained elevated (>/=1 mg/dL) at the next study visit.
Time Frame: Week 52
Population: Intent-to-treat (ITT) population included all participants randomized into the study who received at least one administration of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 50
percentage of participants | 56.0 | 53.1 | 14.0
Statistical Analysis 1: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; The treatment groups were compared using a Cochran-Mantel-Haenszel model adjusted for the stratification factor of starting prednisone dose (less than or equal to [</=] 30 mg/day, greater than [>] 30 mg/day); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Response Rates = 42.00, 99.5% CI 2-sided [18.00 to 66.00]
Statistical Analysis 2: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; The treatment groups were compared using a Cochran-Mantel-Haenszel model adjusted for the stratification factor of starting prednisone dose (</=30 mg/day, >30 mg/day); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Response Rates = 39.06, 99.5% CI 2-sided [12.46 to 65.66]

2. Secondary Outcome: Percentage of Participants in Sustained Remission at Week 52 (Tocilizumab + 26 Weeks Prednisone Taper Versus Placebo + 52 Weeks Prednisone Taper)
Description: Remission was defined as the absence of flare and normalization of the CRP (<1 mg/dL). Sustained remission was defined as the absence of flare following induction of remission within 12 weeks of randomization and maintained up to Week 52. Flare was determined by the investigator and was defined as the recurrence of signs or symptoms of GCA and/or ESR >/=30 mm/hr attributable to GCA. A single CRP elevation (>/=1 mg/dL) was not considered as a sign of flare, unless the CRP remained elevated (>/=1 mg/dL) at the next study visit.
Time Frame: Week 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 51
percentage of participants | 56.0 | 53.1 | 17.6
Statistical Analysis 1: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — The tocilizumab group was to be considered as non-inferior to the placebo group if the lower limit of the two-sided 99.5% confidence interval was >/= -22.5%; Difference in Response Rates = 38.35, 99.5% CI 2-sided [17.89 to 58.81]
Statistical Analysis 3: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Difference in Response Rates = 35.41, 99.5% CI 2-sided [10.41 to 60.41]

3. Secondary Outcome: Time to First GCA Disease Flare
Description: Flare was determined by the investigator and was defined as the recurrence of signs or symptoms of GCA and/or ESR >/=30 mm/hr attributable to GCA. Participants who withdrew from the study prior to Week 52 were censored from the time of withdrawal.
Time Frame: Up to 52 weeks
Population: ITT population
Measure: Median (99% Confidence Interval); unit: days
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 50 | 51
days | NA [NA to NA] — Data could not be calculated due to low number of participants who had an event. | NA [NA to NA] — Data could not be calculated due to low number of participants who had an event. | 165.0 [120.0 to 260.0] | 295.0 [168.0 to NA] — Data could not be calculated due to low number of participants who had an event.
Statistical Analysis 1: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; The treatment groups were compared using a Cox proportional hazards model adjusted for the stratification factor of starting prednisone dose (</=30 mg/day, >30 mg/day); Test type: Superiority or Other; p < 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.23, 99% CI 2-sided [0.11 to 0.46]
Statistical Analysis 2: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0011, Cox proportional hazards model; Hazard Ratio (HR) = 0.39, 99% CI 2-sided [0.18 to 0.82]
Statistical Analysis 3: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, Cox proportional hazards model; Hazard Ratio (HR) = 0.28, 99% CI 2-sided [0.12 to 0.66]
Statistical Analysis 4: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0316, Cox proportional hazards model; Hazard Ratio (HR) = 0.48, 99% CI 2-sided [0.20 to 1.16]

4. Secondary Outcome: Total Cumulative Prednisone Dose
Description: The median total cumulative prednisone dose over the 52 weeks for each treatment group and the corresponding 95% confidence intervals are presented.
Time Frame: Up to 52 weeks
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: milligrams (mg)
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 50 | 51
milligrams (mg) | 1862.00 [1582.0 to 1942.0] | 1862.00 [1568.0 to 2239.5] | 3296.00 [2729.5 to 4023.5] | 3817.50 [2817.5 to 4425.5]
Statistical Analysis 1: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; The treatment groups were compared using a Van Elteren's test stratified by starting prednisone dose (<=30 mg/day, > 30 mg/day); Test type: Superiority or Other; p < 0.0001, Van Elteren's test
Statistical Analysis 2: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Van Elteren's test
Statistical Analysis 3: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; The treatment groups were compared using a Van Elteren's test stratified by starting prednisone dose (<=30mg/day, >30mg/day); Test type: Superiority or Other; p = 0.0003, Van Elteren's test
Statistical Analysis 4: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Van Elteren's test

5. Secondary Outcome: Change From Baseline in Short Form (SF)-36 Questionnaire Score at Week 52
Description: The SF-36 is a standardized questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical Component Score (PCS) and Mental Component Score (MCS). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). A positive change from baseline indicates improvement. No imputation was used for missing data. Data was set to missing for participants who received escape therapy.
Time Frame: Baseline, Week 52
Population: ITT population. Here, 'Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'n' signifies the number of participants evaluable at specified time point for different arms, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 97 | 49 | 48 | 49
units on a scale
  PCS: Baseline (n=97,49,48,49) | 43.10 (9.43) | 40.62 (8.00) | 42.65 (10.87) | 41.12 (9.97)
  PCS: Change at Week 52 (n=59,26,9,18) | 5.37 (7.38) | 2.71 (8.86) | 2.08 (12.11) | -2.80 (6.98)
  MCS: Baseline (n=97,49,48,49) | 42.77 (12.43) | 47.67 (12.59) | 42.73 (12.13) | 40.45 (13.73)
  MCS: Change at Week 52 (n=59,26,9,18) | 8.21 (10.35) | 1.98 (7.17) | 4.99 (7.54) | 2.60 (10.56)
Statistical Analysis 1: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; MCS: Change at Week 52: Repeated measures model used for analysis included the following covariates and interactions: treatment, starting prednisone dose (<=30mg/day, >30mg/day), visit, treatment-by-visit interaction, starting dose-by-visit interaction, baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.8067, Repeated measures model; Difference in Least Square Means = 0.61, 99% CI 2-sided [-5.86 to 7.07]
Statistical Analysis 2: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0252, Repeated measures model; Difference in Least Square Means = 4.44, 99% CI 2-sided [-0.69 to 9.56]
Statistical Analysis 3: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.8374, Repeated measures model; Difference in Least Square Means = -0.56, 99% CI 2-sided [-7.64 to 6.53]
Statistical Analysis 4: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1468, Repeated measures model; Difference in Least Square Means = 3.27, 99% CI 2-sided [-2.59 to 9.14]
Statistical Analysis 5: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; PCS: Change at Week 52: Repeated measures model used for analysis included the following covariates and interactions: treatment, starting prednisone dose (<=30mg/day, >30mg/day), visit, treatment-by-visit interaction, starting dose-by-visit interaction, baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.0570, Repeated measures model; Difference in Least Square Means = 4.38, 99% CI 2-sided [-1.58 to 10.34]
Statistical Analysis 6: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.0024, Repeated measures model; Difference in Least Square Means = 5.59, 99% CI 2-sided [0.86 to 10.32]
Statistical Analysis 7: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.2218, Repeated measures model; Difference in Least Square Means = 3.04, 99% CI 2-sided [-3.43 to 9.51]
Statistical Analysis 8: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.0412, Repeated measures model; Difference in Least Square Means = 4.25, 99% CI 2-sided [-1.14 to 9.64]

6. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Disease Activity Assessed Using Visual Analogue Scale (VAS) at Week 52
Description: Participants assessed their current disease activity on a 0-100 millimeter (mm) VAS, where 0 mm = no disease activity and 100 mm = maximum disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 49 | 51
mm
  Baseline (n=100,49,49,51) | 43.61 (25.66) | 46.65 (25.60) | 35.73 (28.15) | 47.78 (27.80)
  Change at Week 52 (n=60,26,11,18) | -19.68 (33.64) | -22.69 (22.41) | -8.45 (24.81) | -10.00 (35.12)
Statistical Analysis 1: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; Change at Week 52: Repeated measures model used for analysis included the following covariates and interactions: treatment, starting prednisone dose (<=30mg/day, >30mg/day), visit, treatment-by-visit interaction, starting dose-by-visit interaction, baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.0312, Repeated measures model; Difference in Least Square Means = -15.6, 99% CI 2-sided [-34.3 to 3.1]
Statistical Analysis 2: Comparison: Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0476, Repeated measures model; Difference in Least Square Means = -11.8, 99% CI 2-sided [-27.2 to 3.6]
Statistical Analysis 3: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 26 Weeks Prednisone Taper; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0059, Repeated measures model; Difference in Least Square Means = -21.9, 99% CI 2-sided [-42.4 to -1.4]
Statistical Analysis 4: Comparison: Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper vs Part 1: Placebo + 52 Weeks Prednisone Taper; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0081, Repeated measures model; Difference in Least Square Means = -18.2, 99% CI 2-sided [-35.8 to -0.5]

7. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) at Steady State of Tocilizumab
Description: AUCtau is the model-predicted area under the tocilizumab serum concentration versus time curve from time zero to the end of dosing interval. AUCtau is measured in microgram*day per milliliter (mcg*day/mL).
Time Frame: Baseline and Week 16 (Predose [Hour 0], 24, 48, 72, 96, and 120 or 144 hours postdose); Weeks 1, 2, 17, and 18 (Predose [Hour 0])
Population: Pharmacokinetics (PK)-evaluable population included all participants who received at least one tocilizumab injection and had at least one PK sample with detectable results taken at any time during the study.
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49
mcg*day/mL | 499.2 (210.4) | 227.2 (165.4)

8. Secondary Outcome: Maximum Serum Concentration at Steady State (Cmax,ss) of Tocilizumab
Description: Cmax,ss is maximum model-predicted serum steady state concentration of tocilizumab measured in micrograms per milliliter (mcg/mL).
Time Frame: as for outcome 7
Population: PK-evaluable population
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49
mcg/mL | 73 (30.4) | 19.3 (12.8)

9. Secondary Outcome: Minimum Serum Concentration at Steady State (Cmin,ss) of Tocilizumab
Description: Cmin,ss is minimum model-predicted serum steady state concentration of tocilizumab measured in mcg/mL.
Time Frame: as for outcome 7
Population: PK-evaluable population
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49
mcg/mL | 68.1 (29.5) | 11.1 (10.3)

10. Secondary Outcome: Minimum Observed Serum Concentration (Ctrough) of Tocilizumab
Description: Ctrough is minimum observed serum concentration of tocilizumab measured in mcg/mL.
Time Frame: Predose (Hour 0) at Baseline and Week 52
Population: PK-evaluable population. Here, 'Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'n' signifies the number of participants evaluable at specified time point for different arms, respectively.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper
Number analyzed (Participants) | 99 | 48
mcg/mL
  Baseline (n= 99, 48) | 0.07 (0.72) | 0.00 (0.02)
  Week 52 (n= 72, 33) | 67.93 (34.40) | 12.22 (10.02)

11. Secondary Outcome: Serum Interleukin-6 (IL-6) Level
Time Frame: Baseline and Week 52
Population: Safety population. Here, 'n' signifies the number of participants evaluable at specified time point for different arms, respectively.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 50 | 51
picograms per milliliter (pg/mL)
  Baseline (n=91,44,50,47) | 8.79 (10.01) | 16.29 (31.23) | 12.73 (18.04) | 8.31 (9.47)
  Week 52 (n=69,32,28,30) | 65.99 (84.92) | 52.70 (33.10) | 35.96 (149.65) | 10.85 (15.17)

12. Secondary Outcome: Serum Soluble IL-6 Receptor (sIL-6R) Level
Time Frame: Baseline and Week 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 50 | 51
nanograms per milliliter (ng/mL)
  Baseline (n=99,48,50,50) | 51.34 (61.98) | 50.82 (63.51) | 42.07 (11.32) | 40.37 (10.84)
  Week 52 (n=73,33,33,31) | 600.53 (217.52) | 464.30 (153.64) | 76.44 (149.20) | 64.80 (105.13)

13. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
Time Frame: Baseline and Week 52
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: mm/hr
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 50 | 51
mm/hr
  Baseline (n=99,49,50,51) | 19.00 (61.98) [10.00 to 35.00] | 15.00 (63.51) [10.00 to 30.00] | 23.00 (11.32) [9.00 to 36.00] | 20.00 (10.84) [8.00 to 38.00]
  Week 52 (n=76,35,35,33) | 3.00 [2.00 to 5.00] | 5.00 [2.00 to 7.00] | 20.00 [11.00 to 36.00] | 24.00 [10.00 to 37.00]

14. Secondary Outcome: C-Reactive Protein (CRP) Level
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: milligrams per liter (mg/L)
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 100 | 49 | 50 | 51
milligrams per liter (mg/L)
  Baseline (n=100,49,50,51) | 3.67 (61.98) [1.02 to 9.26] | 4.52 (63.51) [1.55 to 9.75] | 3.64 (11.32) [1.20 to 9.59] | 3.56 (10.84) [1.17 to 7.24]
  Week 52 (n=76,35,35,33) | 0.30 [0.20 to 0.59] | 0.33 [0.20 to 0.72] | 4.90 [2.25 to 9.25] | 8.12 [2.02 to 14.40]

15. Secondary Outcome: Percentage of Participants With Anti-Tocilizumab Antibodies
Description: All samples were tested by screening assay, and those samples that were positive were further analyzed by a confirmation assay to confirm specificity. Percentage of participants who has a positive confirmation assay result any time after the initial drug administration with a negative confirmation assay result at baseline was reported.
Time Frame: Baseline up to Week 52
Population: Safety population. Here, 'Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper
Number analyzed (Participants) | 95 | 46 | 49 | 47
percentage of participants | 1.1 | 6.5 | 2.0 | 2.1

ADVERSE EVENTS:
Time Frame: Up to 156 weeks
Description: Safety population
Arm/Group | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper | Part 1: Placebo + 26 Weeks Prednisone Taper | Part 1: Placebo + 52 Weeks Prednisone Taper | Part 2: No Tocilizumab (Placebo in Part 1) | Part 2: No Tocilizumab (Tocilizumab in Part 1) | Part 2: Tocilizumab (Placebo in Part 1) | Part 2: Tocilizumab (Tocilizumab in Part 1)
Serious Adverse Events (participants affected / at risk) | 15/100 | 7/49 | 11/50 | 13/51 | 7/40 | 11/58 | 18/50 | 23/67
Other Adverse Events (participants affected / at risk) | 87/100 | 44/49 | 47/50 | 44/51 | 33/40 | 50/58 | 44/50 | 61/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper (N=100) | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper (N=49) | Part 1: Placebo + 26 Weeks Prednisone Taper (N=50) | Part 1: Placebo + 52 Weeks Prednisone Taper (N=51) | Part 2: No Tocilizumab (Placebo in Part 1) (N=40) | Part 2: No Tocilizumab (Tocilizumab in Part 1) (N=58) | Part 2: Tocilizumab (Placebo in Part 1) (N=50) | Part 2: Tocilizumab (Tocilizumab in Part 1) (N=67)
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 3
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Genital herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry gangrene (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual acuity reduced transiently (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Tocilizumab qw + 26 Weeks Prednisone Taper (N=100) | Part 1: Tocilizumab q2w + 26 Weeks Prednisone Taper (N=49) | Part 1: Placebo + 26 Weeks Prednisone Taper (N=50) | Part 1: Placebo + 52 Weeks Prednisone Taper (N=51) | Part 2: No Tocilizumab (Placebo in Part 1) (N=40) | Part 2: No Tocilizumab (Tocilizumab in Part 1) (N=58) | Part 2: Tocilizumab (Placebo in Part 1) (N=50) | Part 2: Tocilizumab (Tocilizumab in Part 1) (N=67)
Palpitations (Cardiac disorders) | 2 | 2 | 4 | 2 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 3 | 1 | 2 | 2 | 2 | 2
Cataract (Eye disorders) | 5 | 1 | 3 | 4 | 2 | 1 | 3 | 3
Dry eye (Eye disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 4 | 1 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 3 | 8 | 5 | 2 | 2 | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 0 | 2 | 3 | 0
Nausea (Gastrointestinal disorders) | 8 | 2 | 5 | 4 | 1 | 0 | 5 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 3 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 5 | 3 | 5 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 8 | 5 | 8 | 3 | 2 | 2 | 6 | 6
Non-cardiac chest pain (General disorders) | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 16 | 12 | 8 | 6 | 1 | 2 | 5 | 4
Bronchitis (Infections and infestations) | 8 | 4 | 5 | 5 | 4 | 9 | 3 | 9
Conjunctivitis (Infections and infestations) | 4 | 1 | 4 | 1 | 0 | 0 | 4 | 3
Cystitis (Infections and infestations) | 7 | 0 | 2 | 3 | 2 | 3 | 4 | 3
Gastroenteritis (Infections and infestations) | 3 | 4 | 4 | 3 | 0 | 2 | 3 | 4
Nasopharyngitis (Infections and infestations) | 29 | 12 | 9 | 13 | 5 | 13 | 14 | 22
Oral herpes (Infections and infestations) | 4 | 5 | 3 | 2 | 2 | 2 | 1 | 2
Pharyngitis (Infections and infestations) | 4 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 6 | 4 | 2 | 3 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 4 | 1 | 2 | 2 | 1 | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 10 | 6 | 5 | 7 | 1 | 2 | 7 | 2
Urinary tract infection (Infections and infestations) | 10 | 4 | 2 | 4 | 1 | 4 | 10 | 10
Fall (Injury, poisoning and procedural complications) | 7 | 2 | 2 | 2 | 4 | 2 | 2 | 9
Alanine aminotransferase increased (Investigations) | 5 | 2 | 2 | 0 | 0 | 0 | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 1 | 0 | 2 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 8 | 10 | 8 | 7 | 10 | 10 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 7 | 7 | 10 | 3 | 4 | 8 | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6 | 6 | 4 | 0 | 0 | 5 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 6 | 5 | 2 | 4 | 6 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 4 | 4 | 4 | 1 | 0 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 2 | 4 | 2 | 1 | 3 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 2 | 3 | 3 | 1 | 2 | 6 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 5 | 5 | 5 | 1 | 5 | 4 | 7
Dizziness (Nervous system disorders) | 6 | 10 | 6 | 8 | 2 | 0 | 5 | 4
Headache (Nervous system disorders) | 27 | 10 | 16 | 12 | 2 | 8 | 8 | 6
Paraesthesia (Nervous system disorders) | 4 | 2 | 4 | 4 | 0 | 2 | 1 | 5
Tremor (Nervous system disorders) | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 6 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 2 | 3 | 1 | 1 | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 4 | 4 | 0 | 2 | 2 | 4
Sleep disorder (Psychiatric disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 7 | 3 | 2 | 4 | 7 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 3 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 0 | 0 | 0 | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 4 | 8 | 2 | 2 | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 7 | 3 | 5 | 0 | 0 | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 1 | 0 | 2 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 5 | 4 | 2 | 2 | 2 | 0 | 5
Haematoma (Vascular disorders) | 5 | 3 | 3 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 12 | 6 | 4 | 4 | 1 | 7 | 7 | 8
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 4 | 4 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Complement factor C3 decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Complement factor C4 decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 3
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 5
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.